CLINICAL TRIAL: NCT04460209
Title: EP Device Registry
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10316
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Rhythm Disorder
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Standard of Care — Standard of care mapping and/or ablation

SUMMARY:
This study will provide ongoing, high quality data on the safety, performance, and clinical benefits of Abbott's EP devices in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject underwent an electrophysiology imaging (diagnostic procedure) and/or ablation procedure that used one or more Abbott devices covered by this Registry.
* Subject is willing and able to comply with the site's standard of care follow-up schedule.

Exclusion Criteria:

* Subject is currently participating in another clinical investigation that may confound the results of this Registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects of all ages who underwent an electrophysiology (EP) imaging (diagnostic procedure) and/or ablation procedure that used at least one Abbott device covered by this Registry.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a device- and/or procedure-related Serious Adverse Event | 7-days
  that occurred within 7-days of the procedure.
The proportion of procedures that achieved acute success. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sarver, PhD, Study Director — Abbott
Locations (26):
- Austria (2):
  - KH Wiener Neustadt, Wiener Neustadt, Lower Austria
  - A. ö. Krankenhaus der Elisabethinen Linz, Linz, UPR AUS
- FN U sv. Anny v Brno, Brno, Moravia-Silesia, Czechia
- France (3):
  - Pole Sante Republique, Clermont-Ferrand, Auvergne
  - Polyclinique des Fleurs, Ollioules, Provence-Alpes-Azur
  - Clinique Rhône-Durance, Avignon, Provence-Alpes-Côte d'Azur Region
- Germany (3):
  - Deutsches Herzzentrum München des Freistaates Bayern, München, Bavaria
  - Medizinische Einrichtungen der Universität zu Köln, Cologne, North Rhine-Westphalia
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
- Semmelweis University, Budapest, Budapest, Hungary
- India (3):
  - Christian Medical College & Hospital, Vellore, Tmlnadu
  - Max Super Specialty Hospital, New Delhi
  - Sree Chitra Tirunal Institute for Medical Sciences & tech., Trivandrum
- Italy (4):
  - Ospedale San Raffaele, Milan, Lombard
  - Policlinico Universitario A. Gemelli, Roma, Rome
  - Ospedale dell'Angelo, Mestre, Veneto
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Netherlands (3):
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Haga Ziekenhuis Locatie Leyenburg, The Hague, South Holland
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht - Canada
- Portugal (3):
  - Hospital de São João, Porto, Porto District
  - Hospital de Santa Cruz, Carnaxide
  - Hospital Santa Marta, Lisbon
- Spain (3):
  - Hospital General Juan Ramon Jimenez, Huelva, Andalusia
  - Hospital Clínic de Barcelona, Barcelona, Catalon
  - Hospital de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: No